CLINICAL TRIAL: NCT04884880
Title: Prospective, Multicentre, Randomized, Double-blind, Placebo-controlled Clinical Trial of Luo-Fu-Shan Plaster in the Treatment of Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Luo-Fu-Shan Plaster in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director,Devision of Rhenumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020006P4A01
Record Dates: First submitted 2021-04-30; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; External therapy; Herb medicine
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: 180 subjects will be randomized to two parallel groups (90 subjects per group) to receive Luo-Fu-Shan Plaster 10g once daily. Placebo will be administered to individuals randomized to that treatment group in a form identical to the Luo-Fu-Shan Plaster. The first investigational medicinal product dose will be administered the day after the randomization.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luo-Fu-Shan Plaster 10g (Experimental): 10g，once daily，4 weeks
  Interventions: Drug: Luo-Fu-Shan Plaster
- Placebo (Placebo Comparator): 10g，once daily，4 weeks
  Interventions: Drug: The placebo 10g

INTERVENTIONS:
Drug: Luo-Fu-Shan Plaster — Luo-Fu-Shan Plaster 10g，once daily，4 weeks
  Arms: Luo-Fu-Shan Plaster 10g
Drug: The placebo 10g — Placebo 10g，once daily，4 weeks
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the efficacy and safety of Luo-Fu-Shan Plaster in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
The investigators are inspired by Chinese traditonal herb, an therapy for thousands of years, and take its advantage to make Luo-Fu-Shan Plaster in order to get an effective and safe treatment for active RA patients. The study is a multicenter, randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years (time of get informed consent)
* Documented diagnosis of rheumatoid arthritis, as defined by the American Rheumatism Association 1987 Revised Criteria.
* Documented diagnosis of damp-heat syndrome according to Traditional Chinese Medicine.
* If patients are receiving Disease-modifying anti-rheumatic drugs (DMARDs), then the doses should have been kept stable for at least 12 weeks.
* If patients are receiving non-steroidal anti-inflammatory drugs (NSAIDs) or orally Chinese herbal medicine, then the doses should have been kept stable for at least 4 weeks.

Exclusion Criteria:

* Skin allergies or broken skin;
* Taking glucocorticoids,more than 10 mg daily.
* Female patients who are pregnant, breast-feeding or planed to be pregnant;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-05-14 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The changes of Visual Analogue Scale(VAS) pain score | Day 1 to Week 4
  The changes of Visual Analogue Scale(VAS) pain score of global health status, the patient's assessment of pain on a visual analogue scale.
  The score their pain intensity in the most affected joint on a 0-10 cm Visual Analogue Scale Score (VAS), ranging from no pain (0) to extremely pain (10).

SECONDARY OUTCOMES:
The changes of the Disease Activiyu Score (DAS28) | Day 1 to Week 4
  The changes of the Disease Activity Score (DAS28).The score their pain intensity in the most affected joint on a 0-10 cm Disease Activity Score (DAS28), ranging from no pain (0) to extremely pain (10).

OTHER OUTCOMES:
The score of the Health Assessment Questionnaire (HAQ-DI) | Day1 to Week 4
  the patient's assessment of function using a modified version of the Health Assessment Questionnaire (HAQ).The score their level, ranging from no difficuties(0),some difficulties(1),a lot of difficuties(2) to coud not finish(3).
The score of the RA-PRO | Day 1 to Week 4
  the patient's assessment of function using a modified version of the RA-PRO which ranging from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, PhD, Principal Investigator — Guang'anmen Hospital
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No